CLINICAL TRIAL: NCT02744469
Title: Implications of the Population Structure of the Mycobacterium Tuberculosis Complex in Benin for Tuberculosis Presentation, Diagnosis and Outcome
Brief Title: Benin Population Diversity of Tuberculosis and Implications
Acronym: BeniDiT
Status: Completed | Type: Observational
Sponsor: Laboratoire de Référence des Mycobactéries (Other Government)
Collaborators: Direction Générale de la Coopération au Développement, Belgique (Unknown); Institute of Tropical Medicine, Belgium (Other); Universiteit Antwerpen (Other); Laboratoire de Référence des Mycobactéries, Benin republic (Unknown); Centre National Hospitalier Universitaire de Pneumo-Phtisiologie de Cotonou, Benin (Unknown); Centres de Diagnostic et de Traitement de la tuberculose, National Tuberculosis Programme, Benin (Unknown)
Responsible Party: Sponsor
Other Study IDs: LRM-N°030-15/12/2015; CNERS N°030 of 15th/12/2015 (Other: Comité National d'Ethique et de Recherche en Santé du Benin); ITM- N°1040/15 (Other: IRB of Institute of Tropical Medicine Belgium); EC UZA 15/49/532 (Other: University of Antwerp, Belgium; Ethics Committee); Belg registN°:B300201526865 (Other: University of Antwerp, Belgium; Ethics Committee)
Record Dates: First submitted 2016-04-04; First posted 2016-04-20 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; population structure; implications; lineages; spoligotyping; sputum; resistance; culture; diagnostics; outcome; new/retreatment patient
MeSH Terms: conditions — Tuberculosis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputa will be collected at enrolment. Participants will be asked to provide an additional (third) sputum. For the purpose of this study, this sputum will be added to the leftover 2 sputa provided for the routine diagnosis of tuberculosis in order to reach in total at least 5 mL sputum. DNA will be extracted from a part of the sputum for the genotypic characterization Mycobacterium tuberculosis (spoligotype analysis).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- New patients: ''New tuberculosis patients'' are patients just diagnosed for tuberculosis, and who were never treated for tuberculosis or who are treated for less than 1 month. In total, 1192 new patients will be recruited.
  Interventions: Other: No intervention (observational study)
- Retreatment patients: ''Retreatment tuberculosis patients'' are patients just diagnosed for tuberculosis and who were previously treated for tuberculosis (for a duration of 1 month at least). This group includes: patients with treatment relapse, failure and patients who return after default. In total, 298 retreatment patients will be recruited.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study)

SUMMARY:
Tuberculosis is a public health problem caused by a microbe. This microbe may differ from one patient to another. The purpose of this study is to know to which extent, each of these various microbes is involved in tuberculosis disease in Benin. This study will also find out whether the type that affects a patient, depends on patient characteristics and whether the difference affects the outcome of the treatment. Finally the study will also help to find out whether diagnostic tests are reliable for all types of the microbe. This information will be used after the study to inform decision making in order to improve tuberculosis control.

DETAILED DESCRIPTION:
The overall aim of this study is to determine the population structure of Mycobacterium tuberculosis complex in Benin, and implications for tuberculosis presentation, diagnosis and outcome The primary objective is to compare the characteristics of ancestral lineages of Mycobacterium tuberculosis complex, such as M. africanum West African 1 (Lineage 5), with modern M. tuberculosis in Benin.

This study will build on the system of nationwide surveillance already implemented for retreatment patients and recruit in addition a representative random sample of new patients. So for this study sputa from retreatment patients and from a sample of new patients, from the 24 tuberculosis (TB) clinics (Centres de Diagnostic et de Traitement de la Tuberculose) selected all over the country (Benin), will be shipped from TB clinics to the ''Laboratoire de Référence des Mycobactéries'' (LRM), Cotonou (National Reference Laboratory for Mycobacteria, Cotonou) if they consent. All retreatment patients will be recruited into the study and each 4 new patients detected after detection of a retreatment patient will also be recruited into the study.

At enrolment, a questionnaire will be used to collect from consenting participants information such as: Participant place of residence (rural or urban as determined by population density); ethnic group; age; sex; Human Immuno-deficiency Virus (HIV) status; Bacillus Calmette Guerin (BCG) vaccine scar...

Spoligotype analysis will be used to determine the population structure, as it allows the classification of most Mycobacterium tuberculosis complex isolates in lineages, including strains with single or few copies of IS6110.

The external quality evaluation (assurance quality) of the laboratory analyses to be performed at the LRM (National Reference Laboratory for Mycobacteria) in Cotonou, Benin during the study, will be performed by the Institute of Tropical Medicine of Antwerp in Belgium.

ELIGIBILITY:
Inclusion Criteria:

* New or retreatment tuberculosis patients with Acid Fast Bacilli-positive microscopy,
* Diagnosed in a participating TB clinic of Benin,
* Aged ≥15 years (Patients aged less than 15 years old will not be included in this study as acid-fast-bacilli microscopy is rarely positive in children)
* Who has given his/her informed consent (if adult potential participant:≥18 years old) OR who has given his/her assent in addition to the informed consent of his/her legal representative (if potential participant aged 15-<18 years)

Exclusion Criteria:

* Extra-pulmonary TB only,
* New patient who has started taking the TB treatment drugs.
* Retreatment patient who has started taking the TB retreatment drugs.
* Very low sputum quantity (at least 5 milliliters total sputum is acceptable) and potential participant refusing to give more sputum

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There is a National Tuberculosis Program in Benin with a network of 57 TB (tuberculosis) 'diagnosis and treatment centers' (TB clinics). In order to be able to ensure a realistic (cost, time, personnel) strong quality control of data to record on fields in TB clinics, a smaller number of TB clinics where most of Benin TB patients are diagnosed is selected instead of including all the 57 TB clinics. Participants will be recruited from the 4 largest TB clinics of each of Benin's 6 (former) departments (Atlantique/Littoral, Oueme/Plateau, Mono/Couffo, Zou/Collines, Borgou/Alibori, Atacora/Donga), amounting to 24 TB clinics.
Sampling Method: Probability Sample
Enrollment: 1490 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Lineage | At enrollment
  Mycobacterium tuberculosis lineage as determined by the spoligotyping pattern. The lineage will be determined using the specimen collected at participant enrolment. Spoligotyping will be done on sputum, or on culture isolate if failed on sputum and culture is positive.

SECONDARY OUTCOMES:
Spoligotype (family) | At enrollment
  Mycobacterium tuberculosis spoligotype (family) as determined by the spoligotyping pattern. The lineage will be determined using the specimen collected at participant enrolment.
Treatment failure or success as evidenced by microscopy result (for new and retreatment patients) | At Month 6 for new patient; at Month 8 for retreatment patients
  Treatment failure will be ascertained at the end of the treatment period using microscopy for detection of acid-fast bacilli in participant' sputa. Treatment failure or success will be measured using microscopy, only for new and retreatment patients.
Treatment failure or success as evidenced by culture result (for rifampicin resistant patients) | At Month 20 for rifampicin resistant patients
  Treatment failure will be ascertained at the end of the 20 months treatment period by culturing sputa from rifampicin resistant participants.
Relapse ascertainment (by questioning and retrospective check of microscopy evidence in TB clinics) | At Month 18 for new patients; at Month 20 for retreatment patients; at Month 32 for rifampicin resistant patients
  Participants will be called and will be asked whether they have experienced another episode of tuberculosis. This will be retrospectively confirmed in the TB clinic by checking microscopy results for the new episode of tuberculosis.
Chest X-ray findings | At enrollment
  Chest X-ray will be performed in participants to be enrolled in Cotonou and Porto-Novo, the 2 biggest TB clinics and where X-ray is available.
Culture positivity | At enrollment
  Isolation of mycobacteria (in vitro mycobacterial growth) in culture
Phenotypic Drug-resistance or susceptibility | At enrollment (if positive culture)
  Drug resistance as determined using phenotypic drug susceptibility testing on 1st and 2nd line anti-tuberculous drugs
Genotypic resistance to rifampin (GeneXpert) | At enrollment
  Resistance of Mycobacterium tuberculosis to rifampin as determined using the GeneXpert Mtb/Rif test.
(Phenotypic)Type of Mycobacteria (tuberculous or non-tuberculous) | At enrollment (if positive culture)
  Group of Mycobacteria (tuberculous or non-tuberculous) as determined by the result of phenotypic drug sensitivity testing on para-nitro-benzoic acid
(Mpt64's)Type of Mycobacteria (tuberculous or non-tuberculous) | At enrollment (if positive culture)
  Group of Mycobacteria (tuberculous or non-tuberculous) as determined using the Mpt64 antigen test

OTHER OUTCOMES:
Acid-Fast Bacilli microcopy result | 1 Day
  Acid-Fast Bacilli microcopy result on patients' sputa determined using the Ziehl-Neelsen method or the auramine method depending on which of these methods is used at the various tuberculosis clinics where participants will be enrolled.
Acid-Fast Bacilli microcopy on pooled sputum | At enrollment
  Acid-Fast Bacilli microcopy result on the pooled sputum of each participant. The pooled sputum results from the addition of the 2 leftover routine sputa of a participant to the third sputum given after informed consent. This Acid-Fast Bacilli microcopy on pooled sputum will be done after shipment of the pooled sputum to the Reference Laboratory (LRM), using auramine method.
Drug resistance or susceptibility (Novel diagnostic tests) | At enrollment
  Drug resistance pattern for 1st and 2nd lines drugs using novel diagnostic tests.

CONTACTS AND LOCATIONS:
Overall Officials: Dissou Affolabi, MD PhD Prof, Principal Investigator — Laboratoire de Référence des Mycobactéries, Benin; Bouke de Jong, MD PhD Prof, Principal Investigator — Institute of Tropical Medicine, Belgium
Locations (26):
- Institute of Tropical Medicine, Antwerp, Belgium
- Benin (25):
  - Centre de Diagnostic et de Traitement de la Tuberculose de Djougou, Djougou, Atacora/Donga
  - Centre de Diagnostic et de Traitement de la Tuberculose de Matéri, Matéri, Atacora/Donga
  - Centre de Diagnostic et de Traitement de la Tuberculose de Natitingou, Natitingou, Atacora/Donga
  - Centre de Diagnostic et de Traitement de la Tuberculose de Tanguiéta, Tanguiéta, Atacora/Donga
  - Centre de Diagnostic et de Traitement de la tuberculose d'Abomey-Calavi, Abomey-Calavi, Atlantique/Littoral
  - Centre de Diagnostic et de Traitement de la Tuberculose d'Allada, Allada, Atlantique/Littoral
  - Centre National Hospitalier Universitaire de Pneumo-Phtisiologie de Cotonou, Cotonou, Atlantique/Littoral
  - Centre de Diagnostic et de Traitement de la Tuberculose de Ouidah, Ouidah, Atlantique/Littoral
  - Centre de Diagnostic et de Traitement de la Tuberculose de Bembèrèkè HE, Bembèrèkè, Borgou/Alibori
  - Centre de Diagnostic et de Traitement de la Tuberculose de Kandi, Kandi, Borgou/Alibori
  - Centre de Diagnostic et de Traitement de la Tuberculose de Nikki Hopital Sounou-Séro, Nikki, Borgou/Alibori
  - Centre de Diagnostic et de Traitement de la Tuberculose de Parakou CSCom, Parakou, Borgou/Alibori
  - Laboratoire de Référence des Mycobactéries, Cotonou, Littoral Department
  - Centre de Diagnostic et de Traitement de la Tuberculose d'Aplahoué, Aplahoué, Mono/Couffo
  - Centre de Diagnostic et de Traitement de la Tuberculose de Bopa, Bopa, Mono/Couffo
  - Centre de Diagnostic et de Traitement de la Tuberculose de Comè, Comè, Mono/Couffo
  - Centre de Diagnostic et de Traitement de la Tuberculose de Houéyogbé, Péda-Houéyogbé, Mono/Couffo
  - Centre de Diagnostic et de Traitement de la Tuberculose de Avrankou, Avrankou, Oueme/Plateau
  - Centre de Diagnostic et de Traitement de la Tuberculose de Pobè, Pobé, Oueme/Plateau
  - Centre de Pneumo-Phtisiologie d'Akron, Porto-Novo, Oueme/Plateau
  - Centre de Diagnostic et de Traitement de la Tuberculose de Sakété, Sakété, Oueme/Plateau
  - Centre de Diagnostic et de Traitement de la Tuberculose d'Abomey, Abomey, Zou/Collines
  - Centre de Diagnostic et de Traitement de la Tuberculose de Bohicon, Bohicon, Zou/Collines
  - Centre de Diagnostic et de Traitement de la Tuberculose de Dassa-Zoumè, Dassa-Zoumè, Zou/Collines
  - Centre de Diagnostic et de Traitement de la Tuberculose de Zagnanado, Zagnanado, Zou/Collines

REFERENCES:
- [Background] Affolabi D, Anyo G, Faihun F, Sanoussi N, Shamputa IC, Rigouts L, Kestens L, Anagonou S, Portaels F. First molecular epidemiological study of tuberculosis in Benin. Int J Tuberc Lung Dis. 2009 Mar;13(3):317-22. PMID 19275790
- [Background] Brudey K, Driscoll JR, Rigouts L, Prodinger WM, Gori A, Al-Hajoj SA, Allix C, Aristimuno L, Arora J, Baumanis V, Binder L, Cafrune P, Cataldi A, Cheong S, Diel R, Ellermeier C, Evans JT, Fauville-Dufaux M, Ferdinand S, Garcia de Viedma D, Garzelli C, Gazzola L, Gomes HM, Guttierez MC, Hawkey PM, van Helden PD, Kadival GV, Kreiswirth BN, Kremer K, Kubin M, Kulkarni SP, Liens B, Lillebaek T, Ho ML, Martin C, Martin C, Mokrousov I, Narvskaia O, Ngeow YF, Naumann L, Niemann S, Parwati I, Rahim Z, Rasolofo-Razanamparany V, Rasolonavalona T, Rossetti ML, Rusch-Gerdes S, Sajduda A, Samper S, Shemyakin IG, Singh UB, Somoskovi A, Skuce RA, van Soolingen D, Streicher EM, Suffys PN, Tortoli E, Tracevska T, Vincent V, Victor TC, Warren RM, Yap SF, Zaman K, Portaels F, Rastogi N, Sola C. Mycobacterium tuberculosis complex genetic diversity: mining the fourth international spoligotyping database (SpolDB4) for classification, population genetics and epidemiology. BMC Microbiol. 2006 Mar 6;6:23. doi: 10.1186/1471-2180-6-23. PMID 16519816
- [Background] de Jong BC, Antonio M, Gagneux S. Mycobacterium africanum--review of an important cause of human tuberculosis in West Africa. PLoS Negl Trop Dis. 2010 Sep 28;4(9):e744. doi: 10.1371/journal.pntd.0000744. PMID 20927191
- [Background] de Jong BC, Hill PC, Aiken A, Awine T, Antonio M, Adetifa IM, Jackson-Sillah DJ, Fox A, Deriemer K, Gagneux S, Borgdorff MW, McAdam KP, Corrah T, Small PM, Adegbola RA. Progression to active tuberculosis, but not transmission, varies by Mycobacterium tuberculosis lineage in The Gambia. J Infect Dis. 2008 Oct 1;198(7):1037-43. doi: 10.1086/591504. PMID 18702608
- [Background] de Jong BC, Hill PC, Brookes RH, Otu JK, Peterson KL, Small PM, Adegbola RA. Mycobacterium africanum: a new opportunistic pathogen in HIV infection? AIDS. 2005 Oct 14;19(15):1714-5. doi: 10.1097/01.aids.0000185991.54595.41. No abstract available. PMID 16184053
- [Background] Gehre F, Antonio M, Faihun F, Odoun M, Uwizeye C, de Rijk P, de Jong BC, Affolabi D. The first phylogeographic population structure and analysis of transmission dynamics of M. africanum West African 1--combining molecular data from Benin, Nigeria and Sierra Leone. PLoS One. 2013 Oct 15;8(10):e77000. doi: 10.1371/journal.pone.0077000. eCollection 2013. PMID 24143198
- [Background] Affolabi D, Faihun F, Sanoussi N, Anyo G, Shamputa IC, Rigouts L, Kestens L, Anagonou S, Portaels F. Possible outbreak of streptomycin-resistant Mycobacterium tuberculosis Beijing in Benin. Emerg Infect Dis. 2009 Jul;15(7):1123-5. doi: 10.3201/eid1507.080697. PMID 19624936
- [Background] Kamerbeek J, Schouls L, Kolk A, van Agterveld M, van Soolingen D, Kuijper S, Bunschoten A, Molhuizen H, Shaw R, Goyal M, van Embden J. Simultaneous detection and strain differentiation of Mycobacterium tuberculosis for diagnosis and epidemiology. J Clin Microbiol. 1997 Apr;35(4):907-14. doi: 10.1128/jcm.35.4.907-914.1997. PMID 9157152
- [Background] Gagneux S, Small PM. Global phylogeography of Mycobacterium tuberculosis and implications for tuberculosis product development. Lancet Infect Dis. 2007 May;7(5):328-37. doi: 10.1016/S1473-3099(07)70108-1. PMID 17448936
- [Background] Castets M. [Mycobacterium africanum (author's transl)]. Med Trop (Mars). 1979 Mar-Apr;39(2):145-8. French. PMID 91078
- [Background] Parwati I, van Crevel R, van Soolingen D, van der Zanden A. Application of spoligotyping to noncultured Mycobacterium tuberculosis bacteria requires an optimized approach. J Clin Microbiol. 2003 Nov;41(11):5350-1. doi: 10.1128/JCM.41.11.5350-5351.2003. No abstract available. PMID 14605204
- [Background] Asante-Poku A, Yeboah-Manu D, Otchere ID, Aboagye SY, Stucki D, Hattendorf J, Borrell S, Feldmann J, Danso E, Gagneux S. Mycobacterium africanum is associated with patient ethnicity in Ghana. PLoS Negl Trop Dis. 2015 Jan 8;9(1):e3370. doi: 10.1371/journal.pntd.0003370. eCollection 2015 Jan. PMID 25569290
- [Background] Yin X, Zheng L, Lin L, Hu Y, Zheng F, Hu Y, Wang Q. Commercial MPT64-based tests for rapid identification of Mycobacterium tuberculosis complex: a meta-analysis. J Infect. 2013 Nov;67(5):369-77. doi: 10.1016/j.jinf.2013.06.009. Epub 2013 Jun 22. PMID 23796870
- [Derived] Sanoussi CN, de Jong BC, Affolabi D, Meehan CJ, Odoun M, Rigouts L. Storage of Sputum in Cetylpyridinium Chloride, OMNIgene.SPUTUM, and Ethanol Is Compatible with Molecular Tuberculosis Diagnostic Testing. J Clin Microbiol. 2019 Jun 25;57(7):e00275-19. doi: 10.1128/JCM.00275-19. Print 2019 Jul. PMID 31092592
- [Derived] Sanoussi CN, Affolabi D, Rigouts L, Anagonou S, de Jong B. Genotypic characterization directly applied to sputum improves the detection of Mycobacterium africanum West African 1, under-represented in positive cultures. PLoS Negl Trop Dis. 2017 Sep 1;11(9):e0005900. doi: 10.1371/journal.pntd.0005900. eCollection 2017 Sep. PMID 28863143